CLINICAL TRIAL: NCT00086645
Title: Citalopram Treatment in Children With Autism Spectrum Disorders and High Levels of Repetitive Behavior
Brief Title: Citalopram for Children With Autism and Repetitive Behavior (STAART Study 1)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: U54MH066398 (NIH); U54MH066398 (NIH)
Record Dates: First submitted 2004-07-07; First posted 2004-07-13 (Estimated); Last update posted 2017-03-10 (Actual); Status verified 2017-03

CONDITIONS: Autistic Disorder
Keywords: Autism; Asperger Syndrome; Pervasive Developmental Disorder; PDD; Rituals; Compulsions; Stereotypy; Routines; Repetitive behavior; SSRI; Serotonin
MeSH Terms: conditions — Autistic Disorder; Asperger Syndrome; Child Development Disorders, Pervasive; Ceremonial Behavior; Compulsive Behavior; Stereotypic Movement Disorder | interventions — Citalopram

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- citalopram hydrobromide (Experimental): citalopram hydrobromide, up to 20 mg daily
  Interventions: Drug: citalopram hydrobromide
- placebo (Placebo Comparator): placebo, up to equivalent of 20 mg of active comparator daily
  Interventions: Other: placebo

INTERVENTIONS:
Drug: citalopram hydrobromide — 10mg/5ml solution
  Other Names: celexa
  Arms: citalopram hydrobromide
Other: placebo — up to equivalent of 20 mg of active comparator daily
  Arms: placebo

SUMMARY:
This study will determine the efficacy and safety of citalopram compared to placebo in the treatment of children with autism.

DETAILED DESCRIPTION:
For children with autism spectrum disorders (ASD, also known as Pervasive Developmental Disorders - PDDs), repetitive behaviors are common and frequently interfere with functioning in the home as well as in social and educational settings. These behaviors may involve repetitive movements, rigid routines, repetitive play, and even repetitive speech. These behaviors may be associated with high levels of anxiety, severe tantrums. Self-injury can occur when these behaviors and routines are interrupted.

Participants will be randomly assigned to receive citalopram or placebo (administered as liquid), and carefully followed every two weeks. At the end of 12 weeks, children who have responded to treatment will be given the opportunity to continue in the study, with monthly visits, for an additional 24 weeks. Children who received placebo and did not respond to treatment at 12 weeks will be given the opportunity to receive a carefully monitored 12 week course of citalopram.

ELIGIBILITY:
Inclusion Criteria:

* Able to walk
* Diagnosis of Autistic Disorder, Asperger's Disorder, or PDD-NOS
* Have a score greater than or equal to (>) 8 on the sum of items 1A, 2, 3 and 5 of the Compulsions Subscale of the Revised CYBOCS.
* Have a rating of at least moderate behavioral disturbance based on the modified Clinical Global Impression-Severity of Illness score (CGI-S) at the time of screening (See description below).
* Be free of psychotropic medication for at least one month for fluoxetine, two weeks for other SSRIs and neuroleptics, and for 5 days for stimulants prior to baseline ratings.
* Be judged reliable for medication compliance and agree to keep appointments for study contacts and tests as outlined in the protocol (both subject and guardian(s)).

Exclusion Criteria:

* Medical contraindications to therapy with SSRIs
* Prior exposure to citalopram (or escitalopram) of sufficient dose or duration to determine response status
* History of treatment failure to a clinically adequate trial of two select SSRIs
* Diagnosis of Rett's Disorder or Childhood Disintegrative Disorder
* Uncontrolled epilepsy, with a seizure within past 6 months
* Child weighs less than (<) 15 kg at screening contact.
* Pregnancy
* Presence of chronic medical conditions that might interfere with study participation or where study participation would be contraindicated
* Clinically significant abnormal baseline laboratory testing
* History of bipolar disorder or manic episode induced by antidepressant exposure
* Documented need for ongoing psychotropic medications besides study medication (with the exception of stable dose (at least 3 month) anti-convulsants for seizures).
* Concomitant medication that would interfere with participation in the study.
* Recent (< 2 months) initiation of behavior therapy (such as parent training, applied behavior analysis or behavior modification) in a clinic, with a private practitioner or in a school program. Participants who are in an established behavior therapy program (defined as greater than (>) 2 months for clinic or private practitioner or greater than (>) 1 month for school program) can be included in the study. Families will be asked not to initiate any new behavior therapy during the study.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 149 (Actual)
Dates: Start 2004-04; Primary Completion 2006-10 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Clinical Global Improvement | Week 12

SECONDARY OUTCOMES:
Safety Monitoring Uniform Research Form (SMURF) | post-baseline through week 12
Children's Yale-Brown Obsessive-Compulsive Scale (CYBOCS) | Week 12
Repetitive Behavior Scale-Revised (RBS-R) | Week 12
Parent Chief Complaint | Weeks 6 and 12
Aberrant Behavior Checklist | Week 12
Child and Adolescent Symptom Inventory: Anxiety and Depression scales | Week 12
Behavioral Activation | post-baseline through Week 12
Caregiver Strain Questionnaire | Week 12
Vineland | Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Bryan King, MD, Study Chair — University of Washington
Locations (6):
- United States (6):
  - UCLA Neuropsychiatric Institute, Los Angeles, California
  - Yale University, New Haven, Connecticut
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - North Shore - Long Island Jewish Hospital, Great Neck, New York
  - Mount Sinai School of Medicine, New York, New York
  - University of North Carolina Chapel Hill, Chapel Hill, North Carolina

REFERENCES:
- [Derived] Iffland M, Livingstone N, Jorgensen M, Hazell P, Gillies D. Pharmacological intervention for irritability, aggression, and self-injury in autism spectrum disorder (ASD). Cochrane Database Syst Rev. 2023 Oct 9;10(10):CD011769. doi: 10.1002/14651858.CD011769.pub2. PMID 37811711
- [Derived] King BH, Dukes K, Donnelly CL, Sikich L, McCracken JT, Scahill L, Hollander E, Bregman JD, Anagnostou E, Robinson F, Sullivan L, Hirtz D. Baseline factors predicting placebo response to treatment in children and adolescents with autism spectrum disorders: a multisite randomized clinical trial. JAMA Pediatr. 2013 Nov;167(11):1045-52. doi: 10.1001/jamapediatrics.2013.2698. PMID 24061784
- [Derived] King BH, Hollander E, Sikich L, McCracken JT, Scahill L, Bregman JD, Donnelly CL, Anagnostou E, Dukes K, Sullivan L, Hirtz D, Wagner A, Ritz L; STAART Psychopharmacology Network. Lack of efficacy of citalopram in children with autism spectrum disorders and high levels of repetitive behavior: citalopram ineffective in children with autism. Arch Gen Psychiatry. 2009 Jun;66(6):583-90. doi: 10.1001/archgenpsychiatry.2009.30. PMID 19487623